CLINICAL TRIAL: NCT03067961
Title: Investigating the Role of Typhoid Toxin in the Pathogenesis of Enteric Fever: A Double-blinded, Randomised, Outpatient Human Challenge Study.
Brief Title: Investigating Typhoid Fever Pathogenesis
Acronym: TYGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OVG 2016/03
Record Dates: First submitted 2016-12-09; First posted 2017-03-01 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2020-12

CONDITIONS: Salmonella Typhi Infection
Keywords: Enteric fever; Typhoid; Salmonella Typhi; Challenge study; Human model of infection; Typhoid toxin
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wild type S. Typhi Quailes strain (Experimental): Administered by the oral route with sodium bicarbonate at a dose of 1-5x10 4 CFU.
  Interventions: Other: Salmonella Typhi (S. Typhi)
- Quailes typhoid toxin knock-out (Experimental): Administered by the oral route with sodium bicarbonate at a dose of 1-5x10 4 CFU.
  Interventions: Other: Salmonella Typhi (S. Typhi)

INTERVENTIONS:
Other: Salmonella Typhi (S. Typhi) — Investigating the role of typhoid toxin in the pathogenesis of enteric fever

SUMMARY:
Typhoid fever results from infection with a bacterium called Salmonella Typhi and is a major cause of illness worldwide. It is estimated to infect 20-25 million people every year and can affect people of all ages, but is particularly common in young children. The disease is spread through contaminated food and water, and efforts to improve water quality, sanitation and hygiene will likely go a long way to reducing the global burden of disease. Unfortunately, improving access to clean water and sanitation improvements is very costly and difficult to implement on a large scale. Vaccination against typhoid fever is likely to be a cost-effective way of reducing the global disease burden. There are two vaccines currently available against typhoid fever. Whilst these vaccines provide some protection against disease (in the region of 50-70%) these vaccines are less effective in young children, who are the population group at highest risk of disease. In order to develop a new generation of typhoid vaccines it is important to have a more complete understanding of how the bacterium causes disease. In this study, the investigators are aiming to understand more about the Salmonella Typhi bacteria and how it causes disease. In particular, the investigators aim to study the importance of a toxin produced by the typhoid bacteria, called the typhoid toxin. The typhoid toxin has only recently been discovered. It is made only by the typhoid bacteria and closely related bacteria, such as paratyphoid. From studies done in the laboratory, there is evidence that the typhoid toxin is important in causing typhoid disease. It is thought that the typhoid toxin might be important in causing symptoms of typhoid disease, however the exact role of the typhoid toxin during infection in humans hasn't been studied before. Studying this might impact on the design new vaccines against typhoid.

In this study, the investigators will be undertaking a 'challenge' with two strains of the typhoid bacteria (Salmonella Typhi). This involves exposing participants to live Salmonella Typhi under defined circumstances, by asking them to swallow a solution that contains the bacteria. After the challenge the investigators closely monitor participants for a period of at least two weeks and the investigators will then treat participants with antibiotics as soon as they are diagnosed with typhoid disease. The investigators are interested in comparing the response to challenge between two strains of the typhoid bacteria that differ in the production of the typhoid toxin. This process has been undertaken by participants in previous Oxford Vaccine Group studies since 2011.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria to be considered eligible for the study:

* Agree to give informed consent for participation in the study.
* Aged between 18 and 60 years inclusive at time of challenge.
* In good health as determined by medical history, physical examination and clinical judgment of the study team.
* Agree (in the study team's opinion) to comply with all study requirements, including capacity to adhere to good personal hygiene and infection control precautions.
* Agree to allow his or her General Practitioner (and/or Consultant if appropriate), to be notified of participation in the study.
* Agree to allow study staff to contact his or her GP to access the participant's vaccination records and summary of medical history.
* Agree to allow Public Health England to be informed of their participation in the study.
* Agree to give his or her close contacts written information informing them of the participant's involvement in the study and offer them voluntary screening for S. Typhi carriage.
* Agree to have 24-hour contact with study staff during the four weeks post challenge and to be able to ensure that they are contactable by mobile phone for the duration of the challenge period until antibiotic completion.
* Agree to allow the study team to hold the name and 24-hour contact number of a close friend, relative or housemate who will be kept informed of the study participant's whereabouts for the duration of the challenge period (from the time of challenge until completion of antibiotic course). This person will be contacted if study staff are unable to contact the participant.
* Have internet access to allow completion of the e-diary and real-time safety monitoring.
* Agree to avoid antipyretic/anti-inflammatory treatment from the time of challenge (Day 0) until advised by a study doctor or until 14 days after challenge.
* Agree to refrain from donating blood for the duration of the study.
* Agree to provide their National Insurance/Passport number for the purposes of TOPS registration and bank account details for payment of reimbursement expenses.

Exclusion Criteria:

The participant will not be enrolled if any of the following apply:

* History of significant organ/system disease that could interfere with trial conduct or completion. Including, for example, but not restricted to:

  * Cardiovascular disease
  * Respiratory disease
  * Haematological disease
  * Endocrine disorders
  * Renal or bladder disease, including history of renal calculi
  * Biliary tract disease, including biliary colic, asymptomatic gallstones or previous cholecystectomy
  * Gastro-intestinal disease including requirement for antacids, H2-receptor antagonists, proton pump inhibitors or laxatives
  * Neurological disease
  * Metabolic disease
  * Autoimmune disease
  * Psychiatric illness requiring hospitalisation or known or suspected drug and/or alcohol misuse (alcohol misuse defined as an intake exceeding 42 units per week)
  * Infectious disease
* Have any known or suspected impairment of immune function, alteration of immune function, or prior immune exposure that may alter immune function to typhoid resulting from, for example:

  * Congenital or acquired immunodeficiency, including IgA deficiency
  * Human Immunodeficiency Virus infection or symptoms/signs suggestive of an HIV-associated condition
  * Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy.
  * Receipt of immunoglobulin or any blood product transfusion within 3 months of study start.
  * History of cancer (except squamous cell or basal cell carcinoma of the skin and cervical carcinoma in situ).
* Moderate or severe depression or anxiety as classified by the Hospital Anxiety and Depression Score at screening or challenge that is deemed clinically significant by the study doctors .
* Weight less than 50kg .
* Presence of implants or prosthesis.
* Anyone taking long-term medication (e.g. analgesia, anti-inflammatories or antibiotics) that may affect symptom reporting or interpretation of the study results.
* Contraindication to fluoroquinolone or macrolide antibiotics (e.g ciprofloxacin or azithromycin).
* Female participants who are pregnant, lactating or who are unwilling to ensure that they or their partner use effective contraception 30 days prior to challenge and until three negative stool samples have been obtained after completion of antibiotic treatment.
* Full-time, part-time or voluntary occupations involving:

  * Clinical or social work with direct contact with young children (defined as those attending pre-school groups or nursery or aged under 2 years), or
  * Clinical or social work with direct contact with highly susceptible patients or persons in whom typhoid infection would have particularly serious consequences (unless willing to avoid work until demonstrated not to be infected with S. Typhi in accordance with guidance from Public Health England and willing to allow study staff to inform their employer).
* Full time, part time or voluntary occupations involving:

  * Commercial food handling (involving preparing or serving unwrapped foods not subjected to further heating)
* Close household contact with:

  * Young children (defined as those attending pre-school groups, nursery or those aged less than 2 years)
  * Individuals who are immunocompromised.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study period.
* Participants who have participated in another research study involving an investigational product that might affect risk of typhoid infection or compromise the integrity of the study within the 30 days prior to enrolment (e.g. significant volumes of blood already taken in previous study) .
* Detection of any abnormal results from screening investigations (at the clinical discretion of the study team).
* Inability to comply with any of the study requirements (at the discretion of the study staff and the participant's General Practitioner).
* Any other social, psychological or health issues which, in the opinion of the study staff, may

  * put the participant or their contacts at risk because of participation in the study,
  * adversely affect the interpretation of the primary endpoint data,
  * impair the participant's ability to participate in the study.
* Having previously received any typhoid vaccine.
* Having been resident in an enteric fever endemic country for 6 months or more.
* Have previously been diagnosed with laboratory-confirmed typhoid or paratyphoid infection or been given a diagnosis compatible with enteric fever.
* Have participated in previous typhoid or paratyphoid challenge studies (with ingestion of challenge agent).
* Have a prolonged corrected QT interval (>450 milliseconds) on ECG screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical or microbiologically proven typhoid infection | Up to 14 days after challenge dose administered
  The proportion of participants developing clinical or microbiologically proven typhoid infection following oral challenge with 1-5x104 CFU wild type S. Typhi Quailes strain (WT) delivered in a sodium bicarbonate solution, in comparison to challenge with 1-5x104 CFU of a typhoid toxin-deficient isogenic mutant of S. Typhi Quailes strain SB6000 (TN).
  Typhoid fever diagnosis defined as defined as either: i) A positive blood culture for S. Typhi from 72 hours post-challenge or; ii) A positive blood culture for S. Typhi within 72 hours post-challenge, with one or more signs/symptoms of typhoid infection (such as recorded temperature ≥38.0oC) or; (iii) Persistent positive blood cultures (two or more blood cultures taken at least 4 hours apart) for S. Typhi within 72 hours post-challenge or; (iv) Oral temperature ≥38.0oC persisting for 12 hours.

SECONDARY OUTCOMES:
Clinical features following challenge with either wild-type S. Typhi Quailes strain (WT) or typhoid toxin-deficient isogenic mutant S. Typhi Quailes strain SB6000 (TN). | Up to one year after challenge
  Time to onset of symptoms - Time (Days) to first recorded solicited symptoms in the diary card OR first temperature ≥38oC, excluding the first 48 hours following challenge.
Clinical features following challenge with either wild-type (WT) or typhoid toxin-deficient (TN) S. Typhi Quailes strain | Up to one year after challenge
  Duration of illness:Time (Days) from first recorded individual solicited symptoms to complete resolution of individual recorded symptoms in the diary card, excluding the first 48 hours following challenge.
Clinical features following challenge with either wild-type (WT) or typhoid toxin-deficient (TN) S. Typhi Quailes strain | Up to one year after challenge
  Fever clearance time:Time (Hours/Days) from first dose of treatment until temperature ≤37.5°C for a 48 hour period.
Clinical features following challenge with either wild-type (WT) or typhoid toxin-deficient (TN) S. Typhi Quailes strain | Up to one year after challenge
  Symptom severity as measured by: a.The proportion of participants with maximum symptom severity score graded as mild, moderate or severe following challenge; The proportion of participants meeting the criteria for severe enteric fever (Defined as Oral temperature > 40.0oC; Systolic blood pressure < 85 mmHg; Significant lethargy or confusion; Gastrointestinal bleeding; Gastrointestinal perforation; Any grade 4 or above laboratory abnormality, as defined in the study protocol); The proportion of participants reporting the typhoid symptom triad (fever, headache and abdominal pain); The proportion of participants recording one or more severe solicited symptoms following challenge.
  e. Total symptom scores calculated by summing numerical values assigned to the severity of all solicited symptoms between Day 0 to Day 14 (0=not present; 1=mild; 2=moderate; 3=severe);Individual symptom severity scores calculated by summing numerical values assigned to the severity of individual symptoms
Clinical features following challenge with either wild-type (WT) or typhoid toxin-deficient (TN) S. Typhi Quailes strain | Up to one year after challenge
  Time to diagnosis:Time (Hours/Days) from challenge until fulfilment of diagnostic criteria (taken as date/time Gram negative rods are detected in blood culture AND/OR recorded temperature ≥38oC for 12hours)
Microbiological features following challenge with either wild-type (WT) or typhoid toxin-deficient (TN) S. Typhi Quailes strain | Up to one year after challenge
  Time to onset of bacteraemia:(Hours/Days) from challenge until the date/time first positive blood culture collected; Duration of bacteraemia: Time (Hours/Days) from collection of first positive blood culture until date/time of the first negative blood culture and blood cultures are persistently negative;Quantification of bacteraemia at time of diagnosis ( Concentration of bacteria (CFU/ml) in 10ml blood taken at the time of diagnosis using the Wampole™ Isostat® Isolator system (Oxoid Ltd, Basingstoke);Time to onset of stool shedding - Time from challenge (Hours/Days) to the first positive stool culture; Duration of stool shedding - Cumulative number of days where positive stool culture for Salmonella Typhi collected; Pattern of stool shedding - Descriptive
Comparison of haematological and biochemical parameters features following challenge with either wild-type S. Typhi Quailes strain (WT) or typhoid toxin-deficient isogenic mutant S. Typhi Quailes strain SB6000 (TN). | Up to one year after challenge
  •Temporal change and deviation from reference values for the haematological and biochemical parameters below: Total Haemoglobin (g/L) Haemoglobin change from baseline (Hb g/l D0 - Hb g/l D14);Total White Cell Count (x109/l);Platelet counts (x109/l);Neutrophil count (x109/l); Lymphocyte count (x109/l); Monocyte count (x109/l); Eosinophil count (x109/l); Monocyte/Lymphocyte ratio; Urea & Electrolytes (Na, K+, Urea, Creatinine -mmol/l);C-reactive protein (mg/l);Liver function tests (Bilirubin [umol/l], aspartate transaminase (AST IU/l), alkaline phosphatase (ALP IU/l), alanine transaminase (ALT IU/l), Albumin (g/L)
Measures of host immune responses following challenge with either wild-type S. Typhi Quailes strain (WT) or typhoid toxin-deficient isogenic mutant S. Typhi Quailes strain SB6000 (TN). | Up to one year after challenge
  Comparison of the host innate, humoral and cell-mediated responses to challenge with WT and TN strains at baseline (Day 0) and post-challenge time points, with particular reference to, but not limited to: S. Typhi specific antibody concentrations measured by ELISA;Frequency and magnitude of S. Typhi specific antibody-secreting cells as measured by ex-vivo and memory B-cell ELISPOT; Description of lymphocyte populations at baseline and following challenge as measured by flow cytometry and/or CyTOF;Frequency and magnitude of S. Typhi specific cell-mediated immune responses as measured by ELISPOT and flow cytometry and/or CyTOF; Plasma Cytokine concentration
Variation in gene expression in whole blood following challenge with either wild-type S. Typhi Quailes strain (WT) or typhoid toxin-deficient isogenic mutant S. Typhi Quailes strain SB6000 (TN). | Up to one year after challenge
  Comparison of differentially expressed genes using RNASeq on whole blood and/or PBMC samples at baseline (Day 0) and post-challenge time points following challenge with WT and TN strains.
To investigate indirect effects of typhoid-toxin in vivo. | Up to one year after challenge
  Analysis comparing blood and/or urine samples from participants challenged with WT and TN strains, using proteomic and metabolomics based techniques at baseline (Day 0) and post-challenge time points.
Develop methods for direct detection of typhoid toxin in vivo following challenge with wild-type S. Typhi Quailes strain (WT). | Up to one year after challenge
  Exploratory analysis of blood and/or urine and/or faecal samples including use of assays including (but not limited to) mass-spectrometry.
To investigate how the human microbiota, including nasal carriage of Staphylococcus aureus, influences and interacts with a challenge of S. Typhi. | Up to one year after challenge
  Samples of stool, saliva and nasal swabs to measure the constituent microbiological flora by culture and metagenomic studies. • Persistent S. aureus carriage defined as the isolation of S. aureus from at least two samples taken at least one week apart.
To investigate new molecular techniques for detection of S. Typhi in clinical samples. | Up to one year after challenge
  Use of novel methodologies to prepare bacterial DNA/RNA and development of sensitive quantitative and qualitative PCR assays for blood and stool specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, Principal Investigator — Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom, OX3 7LE
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.nature.com/articles/s41591-019-0505-4